CLINICAL TRIAL: NCT01518790
Title: Evaluation of Short Course, Single-dose Polyethylene Glycol (PEG) 3350 Regimen for Colonoscopy Bowel Preparation in Children
Brief Title: Short Course, Single-dose PEG 3350 for Colonoscopy Prep in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 353750
Record Dates: First submitted 2012-01-13; First posted 2012-01-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Colonoscopy
Keywords: PEG 3350; boston bowel preparation scale; colonoscopy cleanout; bowel preparation; miralax; gatorade; cleanout efficacy; Focus of study is efficacy of PEG 3350 cleanout for improving diagnostic yield of colonoscopy.
MeSH Terms: interventions — polyethylene glycol 3350

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Polyethylene glycol 3350 (Experimental)
  Interventions: Drug: polyethylene glycol 3350

INTERVENTIONS:
Drug: polyethylene glycol 3350 — PEG 3350 (238 grams) mixed with 1.9 L (64 oz) of Gatorade, given in 8 oz increments every 15-30 minutes until complete starting at 18:00 on day prior to colonoscopy (max time to completion 6 hours).
  Other Names: Miralax

SUMMARY:
The investigators propose to conduct a prospective study of a widely used bowel preparation regimen (polyethylene glycol 3350 + a sports drink) on pediatric patients who undergo a colonoscopy performed by the pediatric gastroenterology service at WRAMC/WRNMMC between 1 Sep 2010 and 31 Dec 2011. This study will involve the following: determine efficacy of the cleanout, assess tolerability and acceptance of the regimen, determine an appropriate duration to complete the regimen and assess for any electrolyte changes or side effects.

DETAILED DESCRIPTION:
Purpose: It is hoped that by determining acceptability, safety and efficacy of this widely used short course, single-dose bowel preparation regimen, pediatric gastroenterologist can have a standardized bowel preparation for colonoscopy that will be acceptable to pediatric patients and their parents.

Research Design: This study is a prospective medication trial. It will utilize laboratory data to detect any electrolyte changes, a patient questionnaire to assess an acceptable duration, tolerance and side effects of the regimen. Efficacy of the cleanout will be assessed using a published standardized bowel preparation scale by the endoscopist at the completion of the colonoscopy.

Methodology /Technical Approach (including the number of subjects to be studied.): We estimate that 50 patients aged 8-18 years old military dependents who are undergoing a colonoscopy by the Pediatric Gastroenterology service at WRAMC/WRNMMC will be enrolled in the study between 1 Sep 2010 and 31 Dec 2011.

ELIGIBILITY:
Inclusion Criteria:

* Male and female DEERS-eligible dependent military health care beneficiaries age 8 to 18 years old evaluated by Pediatric Gastroenterology service at WRAMC and are scheduled to undergo a colonoscopy between 1 Sep 2010 - 31 Dec 2011 and do not meet exclusion criteria.

Exclusion Criteria:

* Age less than 8 years or greater than 18 at time of procedure
* Colonic surgery including hemicolectomy, colectomy, ileostomy, or multiple abdominal surgeries.
* Oral aversion or other feeding disorder.
* Inability to drink large amount of liquids.
* Aspiration risk.
* Renal disease or pre-cleanout electrolytes outside normal range.
* Significant cardiovascular disease.
* Allergy to food coloring or polyethylene glycol 3350.
* Inpatient or emergency colonoscopy.
* Current nasogastric tube in place.
* Known Pregnancy. Urine pregnancy test will only be completed on day of colonoscopy for all females age 14 and older per current standard anesthesia protocols. There have been no known reported animal or human studies that report the fetal effects of using polyethylene glycol. Per FDA, it is labeled as a category C drug in pregnancy. However, two studies , have reported successful treatment of constipation during pregnancy using polyethylene glycol solutions and did not find any significant effects or safety issues

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of Cleanout | At the end of the colonoscopy within 10-18 hours of completing the cleanout
  Efficacy of cleanout utilizing Boston bowel preparation scale, completed by endoscopy fellow and staff at the end of the colonoscopy done within 10-18 hours after completion of the cleanout.

SECONDARY OUTCOMES:
Electrolyte changes assessing basic metabolic profiles pre/post cleanout | 30 days prior to 1 day after cleanout
  BMP will be obtain within 30 days of cleanout and on the day of the colonoscopy at the time of IV insertion for anesthesia.
Patient/parent satisfaction/tolerability/side effects utilizing questionnaire | 1 day after cleanout
  Parents or patient fill out questionnaire on day of the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mazen I Abbas, DO, MPH, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Abbas MI, Nylund CM, Bruch CJ, Nazareno LG, Rogers PL. Prospective evaluation of 1-day polyethylene glycol-3350 bowel preparation regimen in children. J Pediatr Gastroenterol Nutr. 2013 Feb;56(2):220-4. doi: 10.1097/MPG.0b013e31826630fc. PMID 22744195